CLINICAL TRIAL: NCT05243316
Title: Risk of 24 Hour-pneumothorax After Chest Tube Removal With and Without Chest Tube Clamping in Patients With Pleural Pathology at the National Institute of Respiratory Diseases
Brief Title: Risk of Pneumothorax With and Without Chest Tube Clamping in Patients With Pleural Pathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C58-21
Record Dates: First submitted 2022-01-31; First posted 2022-02-17 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2022-02

CONDITIONS: Pneumothorax; Chest Tube; Pleural Diseases
Keywords: Chest tube; Pneumothorax; Pleural Diseases
MeSH Terms: conditions — Pneumothorax; Pleural Diseases | interventions — Constriction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Randomizing will be masked, as well as data analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with clamping of the chest tube (Active Comparator): Patients with 6hour clamping prior to removal
  Interventions: Procedure: Clamping
- Patients without clamping of the chest tube (Sham Comparator): Patients will have chest tube removed immediately
  Interventions: Procedure: Non Clampling

INTERVENTIONS:
Procedure: Clamping — There will be a randomized selection of patients who will have a clamping of the chest tube 6 hours prior to chest tube removal.
  Arms: Patients with clamping of the chest tube
Procedure: Non Clampling — There will be a randomized selection of patients who wont have chest tube clamping 6 hours prior to chest tube removal.
  Arms: Patients without clamping of the chest tube

SUMMARY:
Through this randomized controlled clinical trial, we aim to identify whether there is a difference in the incidence of 24 hour pneumothorax after chest tube removal, in two blindly randomized groups of patients: The first group with chest tube clamping 6 hours prior to removal, and the second group there will be no chest tube clamping.

The data will be prospectively collected from patient records from the National Institute of Respiratory Diseases Ismael Cosío Villegas.

DETAILED DESCRIPTION:
Patients with an indication of chest tube removal will be randomized to two possible arms: clamping (for 6 hours before removal) or not clamping (immediate removal).

Incidence of 24hour pneumothorax after chest tube removal will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 years and more.
* Patients hospitalized in the National Institute of Respiratory Diseases.
* Patients who had a chest tube placement during their stay at the hospital, by any cause.

Exclusion Criteria:

* Patients who refuse to sign the informed consent and who refuse to participate in the study.
* Patients who die before randomization.
* Patients who gets chest tube removal before being randomized.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Incidence of pneumothorax after chest tube removal with chest tube clamping | After 24 hours of procedure
  Cases of pneumothorax after chest tube removal despite clamping
Incidence of pneumothorax after chest tube removal without chest tube clamping | After 24 hours of procedure
  Cases of pneumothorax after chest tube removal despite clamping

SECONDARY OUTCOMES:
Hospital days of stay | Through study completion, an average of 1 month
  Hospital days of stay

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Rodriguez, Doctor, Study Director — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- National Institute of Respiratory Diseases, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Database will be available once the protocol is complete
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Once completed for one year
Access Criteria: Free access